CLINICAL TRIAL: NCT01767025
Title: The Influence of Oxytocin on Automatic Imitation Behaviour in Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2012/550
Record Dates: First submitted 2013-01-10; First posted 2013-01-11 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: Influence; oxytocin; automatic imitation; behaviour; volunteers
MeSH Terms: conditions — Behavior | interventions — Oxytocin; Seawater

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin (Experimental): Oxytocin 24 IU (3 puffs) per nostril
  Interventions: Drug: Oxytocin
- Sea water (Placebo Comparator): Sea water 3 puffs per nostril
  Interventions: Drug: Sea water

INTERVENTIONS:
Drug: Oxytocin
  Arms: Oxytocin
Drug: Sea water
  Arms: Sea water

SUMMARY:
In this study, the influence of oxytocin on automatic imitation behaviour is investigated. Healthy adults will be administered with either oxytocin or a placebo, and will perform an imitation-inhibition task (as a measure of automatic imitation behaviour). To determine the specificity of the oxytocin effect, an unrelated cognitive task (Stroop task) will also be presented.

ELIGIBILITY:
Inclusion Criteria:

* Male
* non-smoker

Exclusion Criteria:

* no pacemaker, deep brain stimulation electrodes or other stimulation devices
* normal neurological history (no brain operations, migraine, epilepsy, alcoholism
* no epilepsy in family
* no chronic disease(s) that require constant medication (asthma, hypertension, diabetes)
* no medication 24h prior to experiment
* no alcohol or caffeine 2h prior to experiment
* no sleep deprivation 24h prior to experiment

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the automatic imitation behaviour 45 minutes after drug administration | 120 minutes
  Since the effects of oxytocin are only visible after 45 minutes, participants will have to wait 45 minutes before starting the experimental tasks. In the meantime, they will be given an unrelated cognitive-emotional filler task which will last ± 30 minutes. Afterwards, they will perform two experimental tasks: an imitation-inhibition task and a cognitive control task (Stroop task).

CONTACTS AND LOCATIONS:
Overall Officials: Guy T'Sjoen, MD, PhD, Principal Investigator — Ghent University, Faculty of Endrocrinology
Locations (1):
- Ghent University, Faculty of Psychology and Educational Sciences, Ghent, Belgium